CLINICAL TRIAL: NCT07174089
Title: New AI-based Technologies for Even Safer and More Precise Nuclear Medicine
Brief Title: New AI-based Technologies in Nuclear Medicine
Acronym: AI-basedMedNuc
Status: Recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 267/2022/SPER/IRCCSRE
Record Dates: First submitted 2025-09-04; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Patients Undergoing PET/CT Investigation or Nuclear Medicine Therapy
Keywords: extravasation; SUV; radioligand therapy; radiopharmaceutical; dosimetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing radiotherapy: The individuals studied will all be patients administered with radiopharmaceuticals for diagnostic and therapy purposes (aged between 18 and 90).
  Interventions: Other: RadEye SPRD-ER device: spectrometric radiation detector capable of detecting gamma radiation.

INTERVENTIONS:
Other: RadEye SPRD-ER device: spectrometric radiation detector capable of detecting gamma radiation. — Acquisition of data during the infusion of PET radiotracers and the administration of α and β emitting radiopharmaceuticals for therapy.

SUMMARY:
The study aims to identify and predict radiopharmaceutical extravasation events using new semi-quantitative parameters and machine learning models. It involves dose rate measurements to develop metrics for real-time monitoring. It also investigates the correlation between extravasation and SUV correction in PET/CT diagnostics, providing an estimate of the correction factor necessary for accurate SUV evaluation in case of an extravasation event.

DETAILED DESCRIPTION:
This is a descriptive, observational, non-profit study aimed at detecting and predicting extravasation events during the administration of radiopharmaceuticals for diagnostic and therapeutic purposes in nuclear medicine. Extravasation can lead to local tissue damage and compromise the accuracy of semi-quantitative imaging parameters such as the Standardized Uptake Value (SUV), widely used in PET/CT for diagnosis, staging, and therapy response evaluation. Literature reports that extravasation may cause a 21-50% change in SUV, potentially leading to incorrect assessment of tumor response.

The study will use a CE-marked portable spectroscopic personal radiation detector (RadEye SPRD-ER, Thermo Fisher Scientific™), already validated in a previous Ethics Committee-approved study, to record dose-rate (DR) curves during radiopharmaceutical injections. Using these data, new dosimetric metrics will be developed to characterize correct, abnormal, and extravasation events. Machine learning (ML) algorithms will be trained on patient clinical data, injection metrics, and DR curves to classify injection events in real time and to estimate correction factors for SUV quantification. Monte Carlo simulations (MCNP code, anthropomorphic phantoms, and reconstructed patient geometries) will be performed to evaluate absorbed dose distributions in extravascular regions.

The project is structured into three phases:

Phase 1 (Data Acquisition & Analysis): Real-time monitoring with RadEye SPRD-ER, extraction of quantitative metrics (DRmax, DRmean, Δp, t*, Δt), development of ML classifiers and regression models for SUV correction.

Phase 2 (Monte Carlo Simulations): Activity and dose calibration, dose distribution modeling in extravascular tissues.

Phase 3 (Dissemination): Scientific publications and presentation of results at international conferences.

This study has the potential to improve safety, diagnostic reliability, and accuracy of radiopharmaceutical administrations by introducing predictive monitoring and real-time correction of quantitative imaging parameters.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing PET/CT scans or therapeutic treatments with radiopharmaceuticals labelled with alpha or beta emitting nuclides

Exclusion Criteria:

* patients whose clinical or psychological conditions do not allow for their involvement

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing standard-of-care nuclear medicine procedures (PET/CT or therapeutic α/β radiopharmaceutical administrations).
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Characterization of new semi-quantitative metrics to detect extravasation events | During and immediately after radiopharmaceutical injection
  Identification and validation of quantitative parameters derived from dose-rate (DR) curves capable of reliably distinguishing between normal injection, abnormal venous retention, and extravasation events. Metrics will be applicable to both therapeutic radiopharmaceuticals (α and β emitters) and diagnostic radiotracers (e.g., PET/CT)

SECONDARY OUTCOMES:
Correlation between extravasation severity and SUV alterations in nuclear medicine diagnostics | within 90 minutes after radiopharmaceutical administration
  Identification and quantification of the relationship between the extent of radiopharmaceutical extravasation and changes in Standardized Uptake Value (SUV) in diagnostic imaging. This analysis will be performed using Monte Carlo simulations and OLINDA software for activity estimation and dosimetric calibration. Patient-specific imaging data (CT, PET) will be used to model extravasation events and evaluate their impact on SUV quantification.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, Italy

REFERENCES:
- [Background] Wilson S, Osborne D, Long M, Knowland J, Fisher DR. Practical Tools for Patient-specific Characterization and Dosimetry of Radiopharmaceutical Extravasation. Health Phys. 2022 Nov 1;123(5):343-347. doi: 10.1097/HP.0000000000001600. Epub 2022 Jul 15. PMID 35838538
- [Background] Iori M, Grassi E, Piergallini L, Meglioli G, Botti A, Sceni G, Cucurachi N, Verzellesi L, Finocchiaro D, Versari A, Fraboni B, Fioroni F. Safety injections of nuclear medicine radiotracers: towards a new modality for a real-time detection of extravasation events and 18F-FDG SUV data correction. EJNMMI Phys. 2023 May 23;10(1):31. doi: 10.1186/s40658-023-00556-5. PMID 37221434
- [Background] Tylski P, Pina-Jomir G, Bournaud-Salinas C, Jalade P. Tissue dose estimation after extravasation of 177Lu-DOTATATE. EJNMMI Phys. 2021 Mar 31;8(1):33. doi: 10.1186/s40658-021-00378-3. PMID 33788043
- [Background] Kiser JW, Benefield T, Lattanze RK, Ryan KA, Crowley J. Assessing and Reducing Positron Emission Tomography/Computed Tomography Radiotracer Infiltrations: Lessons in Quality Improvement and Sustainability. JCO Oncol Pract. 2020 Jul;16(7):e636-e640. doi: 10.1200/JOP.19.00302. Epub 2020 Feb 11. PMID 32045542
- [Background] Williams JM, Arlinghaus LR, Rani SD, Shone MD, Abramson VG, Pendyala P, Chakravarthy AB, Gorge WJ, Knowland JG, Lattanze RK, Perrin SR, Scarantino CW, Townsend DW, Abramson RG, Yankeelov TE. Towards real-time topical detection and characterization of FDG dose infiltration prior to PET imaging. Eur J Nucl Med Mol Imaging. 2016 Dec;43(13):2374-2380. doi: 10.1007/s00259-016-3477-3. Epub 2016 Aug 25. PMID 27557845
- [Background] Osborne D, Lattanze R, Knowland J, Bryant TE, Barvi I, Fu Y, Kiser JW. The Scientific and Clinical Case for Reviewing Diagnostic Radiopharmaceutical Extravasation Long-Standing Assumptions. Front Med (Lausanne). 2021 Jun 28;8:684157. doi: 10.3389/fmed.2021.684157. eCollection 2021. PMID 34262915
- [Background] Bilgic S. FDG Extravasation in PET/CT Imaging: A Visual Grading Approach Based on Clinical Observations. J Med Imaging Radiat Oncol. 2025 Sep;69(6):617-625. doi: 10.1111/1754-9485.13876. Epub 2025 Jul 2. PMID 40600568
- [Background] van der Pol J, Voo S, Bucerius J, Mottaghy FM. Consequences of radiopharmaceutical extravasation and therapeutic interventions: a systematic review. Eur J Nucl Med Mol Imaging. 2017 Jul;44(7):1234-1243. doi: 10.1007/s00259-017-3675-7. Epub 2017 Mar 16. PMID 28303300